CLINICAL TRIAL: NCT05444023
Title: Comparison of Suturing Technique Types on Pubocervical Fascia at Colporrhaphy Anterior for Cystocele Repair
Brief Title: Comparison of Suturing Technique Types on Pubocervical Fascia at Colpographhy Anterior for Cystocele Repair
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kanuni Sultan Suleyman Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Ozan Karadeniz, Principal investigator, Kanuni Sultan Suleyman Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KanuniSSEAH
Record Dates: First submitted 2022-06-24; First posted 2022-07-05 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-03

CONDITIONS: Pelvic Organ Prolapse
Keywords: anterior colporrhaphy; pubocervical fascia; suturing technique; cycstocele; pelvic organ prolapse
MeSH Terms: conditions — Pelvic Organ Prolapse

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Transverse separated suturing technique (Experimental): During pubocervical fascia reconstruction, the surgeon will perform suturing at the transverse plane with an intermittent stitching technique.
  Interventions: Procedure: Pubocervical fascia reconstruction
- circular continue suturing technique (Active Comparator): During pubocervical fascia reconstruction, the surgeon will perform a continuous stitching technique which includes the lateral parts of the anterior compartment defect.
  Interventions: Procedure: Pubocervical fascia reconstruction

INTERVENTIONS:
Procedure: Pubocervical fascia reconstruction — Suturing type techniques on pubocervical fascia reconstruction at anterior compartment defects.

SUMMARY:
Anterior colporrhaphy is the commonly performed surgery for pelvic organ prolapse. However the success rates of native tissue repair techniques for anterior vaginal prolapse range from %30-%70. According to a systematic review of the anterior colporrhaphy technique, there was no ideal procedure or guideline for gynecologists to perform. The investigators tried to compare pubocervical fascia suturing techniques with the ideal procedure type by determining step by step all parts of the surgery including the anesthesia type. The aim of the study will be to compare the pubocervical fascia reconstruction techniques in the management of anterior compartment defects (POP-Q >2) at 1 year and yearly up to 2 years.

DETAILED DESCRIPTION:
Primary and secondary endpoints:

Primary outcome measures will be the subjective cure of prolapse ("absence or presence of a bulge in the vagina"), objective success with anatomic absence of advanced prolapse at POP-Q sites Ba, C and Bp defined as less than 1 cm individually and as a total.

Secondary outcome measures include all other parameters such as perioperative outcomes, patient satisfaction, quality of life outcomes, complications, scores on questionnaires, and reoperations.

The study protocol will be submitted to the institutional review boards of every participating study site and written informed consent will be obtained from all participants on enrolment.

Project design: The investigators will perform an international singlecentre single-blind randomized controlled trial by participating in our tertiary referral hospital.

ELIGIBILITY:
Inclusion Criteria:

* Women with symptomatic stage 2 or greater (point C -1 or more pelvic organ prolapse quantification POP-Q) cystocele
* Women aged between 18-75 years of age

Exclusion Criteria:

* Women not eligible for surgery for medical or anesthesiological reasons
* Inability to comprehend questionnaires
* Inability to give informed consent
* Inability to return for a review
* Prior anterior compartment repair with or without mesh
* Severe cardiovascular or respiratory disease
* Women who don't want anterior compartment repair
* Pregnancy
* Age <18 years

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-11-15 (Actual); Primary Completion 2023-11-15 (Actual); Study Completion 2024-03-03 (Actual)

PRIMARY OUTCOMES:
Subjective cure rate of prolapse | Time Frame: 12 months after intervention
  Provided by the patient's feeling of the "Absence of a bulge in the vagina"
Objective success | Time Frame: 12 months after intervention
  Defined as anatomic absence of advanced prolapse at POP-Q sites Ba, C and Bp defined as less than 1 cm individually and as a total

SECONDARY OUTCOMES:
Prolapse-related Quality of life | Time Frame: 12 months after intervention
  This will be assessed using a validated questionnaire (Prolapse Quality of Life questionnaire P-QoL) The questionnaire contains 9 domains. Each answer of the patient will have values that range between 1 to 4 or 1 to 5 for the 1st question only). (1 very good 4/5 very poor). There is no overall score. A symptomatic woman might have only one domain impaired and another one might have all domains impaired. We consider both of them symptomatic but in different or same aspects of quality of life. To differentiate different domains, it is important for the decision of our surgery (we will be careful in shortening and narrowing a vagina of a woman who had only a preoperative high (impaired) Personal relationships domain score and other domains in the normal range).
  This will also help us in the follow up visits.
Failure (%) | Time Frame: 12 months after intervention
  Recurrence rate
Complications | Time Frame: 12 months after intervention
  İnjury ( bowel, intestinal, blood vessel injuries)
Pelvic Organ Prolapse/Urinary Incontinence Sexual Questionnaire (PISQ-12) | Time Frame: 12 months after intervention
  The PISQ-12 is a self-adminestered questionnaire that evaluates sexual function of women with pelvic organ prolapse or urinary incontinence. The questionnaire has 12 items. Other than the first 4 questions that are scored from 4 to 0, all questions are scored from 0 to 4. The total score is calculated with totaling the score of each question. The maximum score is 48. Higher scores show good sexual functioning of women.
Incontinence Impact Questionnaire (IIQ-7) | Time Frame: 12 months after intervention
  evaluating the impact of urinary incontinence
Pelvic Floor Distress Inventory (PFDI - 20) | Time Frame: 12 months after intervention
  evaluating the bowel, bladder, or pelvic symptoms

CONTACTS AND LOCATIONS:
Locations (1):
- Kanuni Sultan Suleyman Training and Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided